CLINICAL TRIAL: NCT02067533
Title: Flexion Versus Extension Soft Tissue Repair in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amin Nemati, Orthopedic surgery resident,Orthopedic department,Alzahra hospital,Isfahan University of Medical Sciences,Isfahan,Iran, Isfahan University of Medical Sciences
Other Study IDs: 390187
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Total Knee Arthroplasty(TKA); Total Knee Replacement

ARMS (2):
- flexion position (Experimental)
  Interventions: Procedure: soft tissue repair in flexion position
- extension position (Experimental)
  Interventions: Procedure: soft tissue repair in extension position

INTERVENTIONS:
Procedure: soft tissue repair in flexion position
  Arms: flexion position
Procedure: soft tissue repair in extension position
  Arms: extension position

SUMMARY:
The purpose of the present study is to determine the influence of position of soft tissue repair (flexion versus extension) in post operative range of motion(ROM) and functional outcome in patients who underwent primary total knee arthroplasty (TKA).

ELIGIBILITY:
Inclusion Criteria:

* were individuals with osteoarthritis indicated for primary Total Knee Arthroplasty

Exclusion Criteria:

* previous fracture in thigh
* previous fracture in leg
* previous high tibial osteotomy

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Primary Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vice Chancellery for Research of Isfahan University of Medical Sciences, Isfahan, Iran, Isfahan, Isfahan, Iran

RESULTS

PARTICIPANT FLOW:
Groups:
- Flexion Position: soft tissue repair in flexion position
- Extension Position: soft tissue repair in extension position
Period: Overall Study
Arm/Group | Flexion Position | Extension Position
Started | 45 | 46
Completed | 41 | 44
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flexion Position | Extension Position | Total
Number analyzed (Participants) | 45 | 46 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (8.6) | 67.5 (7.6) | 67.14 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 40 | 74
  Male | 11 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Knee Range of Motion (ROM)
Description: in all patients ROM is measure 1 year after knee surgery by one of the study investigator using goniometer.
Time Frame: 1 year after total knee arthroplasty
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Flexion Position | Extension Position
Number analyzed (Participants) | 41 | 44
degree | 119 (6.8) | 120 (5.4)

ADVERSE EVENTS:
Arm/Group | Flexion Position | Extension Position
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/44
Other Adverse Events (participants affected / at risk) | 0/41 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No